CLINICAL TRIAL: NCT06148935
Title: Post-marketing Surveillance Study for Verquvo (Vericiguat) in Korean Heart Failure Patients With Reduced Ejection Fraction
Brief Title: An Observational Study to Learn More About the Use of Vericiguat in Korean People With Chronic Heart Failure With Reduced Ejection Fraction (HFrEF) in Real-world Setting
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22013
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — vericiguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Korean adult participants with HFrEF: Korean heart failure participants with reduced ejection fraction (HFrEF) who are prescribed Verquvo (Vericiguat) for an approved indication by the Ministry of Food and Drug Safety (MFDS) in Korea
  Interventions: Drug: Vericiguat (Verquvo, BAY1021189)

INTERVENTIONS:
Drug: Vericiguat (Verquvo, BAY1021189) — Following the manner of observational study, no intervention will be provided in the study. Participants follow locally approved label, without interference by the study initiator or study protocol

SUMMARY:
This is an observational study in which only data are collected from participants receiving their usual treatment. The study is done in people with chronic heart failure with reduced ejection fraction (HFrEF). HFrEF is a long-term condition in which the heart does not pump blood as well as it should. Blood and fluid may collect in the lungs, blood vessels, and tissues causing shortness of breath or tiredness. Over time, heart failure can lead to other serious medical conditions that may result in hospital stays and death.

The study treatment vericiguat works by increasing the activity of an enzyme called soluble guanylate cyclase (sGC). sGC helps to regulate the heart and blood circulation. Vericiguat has already been studied in previous clinical studies and is available for doctors to prescribe to people with heart failure. This study will collect important data from real-world setting in Korea. The participants of this study are people with HFrEF who will receive vericiguat as prescribed by their doctors according to the approved product information

The main purpose of this study is to learn more about how safe vericiguat is in the participants. To do this, researchers will collect data on all medical problems (also called adverse events) that the participants have during the study. Doctors keep track of all adverse events, even if they do not think they might be related to the study treatment.

Further, researchers will collect data on how well vericiguat works and treatment patterns in the participants. For this, the following information will be collected:

* occurrence of death due to heart and circulatory events
* hospital stays due to heart conditions (failure)
* dose levels of vericiguat and duration of treatment

The data for this study will come from medical records and visits that take place in routine practice. Participants will be treated with vericiguat and observed up to 12 months or until death or they leave the study, whatever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 19 years or older
* Chronic HF (NYHA functional class II, III, or IV) Reduced left ventricular ejection fraction (< 45%) within 12 months before enrollment
* Worsening of heart failure (hospitalized within 6 months before enrollment or intravenous diuretic therapy without hospitalization within 3 months)
* Participants who have been prescribed Verquvo (Vericiguat) as per locally approved label and didn't receive Verquvo (Vericiguat) therapy previously.
* Written informed consent from subject or legal representative; assent from subject when appropriate

Exclusion Criteria:

* Contraindication according to the local authorized label (including known hypersensitivity to the drug substance or any of its components, pregnancy)
* Participants participating in an investigational program with interventions outside of routine clinical practice

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female and male participants with a diagnosis of heart failure with reduced ejection fraction (HFrEF) will be enrolled after the decision for treatment with Verquvo (Vericiguat) has been made by the investigator´s discretion.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs), serious adverse events (SAEs), adverse drug reactions (ADRs), serious adverse drug reactions (SADRs), unexpected adverse events (unexpected AEs) and unexpected adverse drug reactions (unexpected ADRs) | From the date first administration of Verquvo (Vericiguat) to 14 days after the end of the treatment period, up to 12 months for each participant.

SECONDARY OUTCOMES:
Occurrence of the composite of cardiovascular (CV) death or first hospitalization due to heart failure (HF) | From initial visit to final visit, up to 12 months for each participant
Occurrence of CV death | From initial visit to final visit, up to 12 months for each participant
Occurrence of HF hospitalization | From initial visit to final visit, up to 12 months for each participant
Time to reach different dose levels of Verquvo (Vericiguat) during initial titration | From initial visit to final visit, up to 12 months for each participant
Relative time on different dose levels of Verquvo (Vericiguat) during follow-up | From first follow-up visit to final visit, up to 11 months for each participant

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, South Korea

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.